CLINICAL TRIAL: NCT05601492
Title: Adherence to Otezla in Patients With Mild Psoriasis
Brief Title: Adherence to Otezla
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Terminated IRB approval 6/26/2024, study was never initiated or activated
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: IRB00088889
Record Dates: First submitted 2022-10-13; First posted 2022-11-01 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — apremilast

STUDY DESIGN:
Intervention Model Description: Randomization 1:1:1
Who Masked: Participant
Masking Description: The participant will not know that the electronic cap adapter is actually recording the opening of the medication bottle.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Arm 1 - Standard of Care (Active Comparator): Participant will be given the medication with an electronic monitoring cap attached and a return appointment for a standard of care regular visit
  Interventions: Drug: Otezla - Standard Care; Behavioral: Reminder Text Intervention with apremilast; Behavioral: Extended Consultation for apremilast
- Arm 2 - Reminder text (Experimental): Participant will be given the medication with an electronic monitoring cap attached and receive weekly electronic text/email-based reporting intervention that is designed to promote better adherence to treatment (to help assure that the study have subjects who have excellent adherence. Having patients report their progress on a regular basis promotes better treatment adherence, perhaps by creating the same sense of accountability promoted by regular office visits
  Interventions: Behavioral: Reminder Text Intervention with apremilast
- Arm 3 - Initial patient consult (Experimental): Participant will be given the medication with an electronic monitoring cap attached and will receive an initial patient consultation intervention, which will focus on the prescribed medication education and setting expectations of what to anticipate with usage of the medication
  Interventions: Behavioral: Extended Consultation for apremilast

INTERVENTIONS:
Drug: Otezla - Standard Care — The participant will be given their medication with the electronic adapter cap on it and asked to return for the follow-up visit
  Other Names: Apremilast
  Arms: Arm 1 - Standard of Care
Behavioral: Reminder Text Intervention with apremilast — Participants will receive a weekly electronic text/email-based intervention that is designed to promote better adherence to treatment in addition to receiving their medication with the electronic adapter cap on it.
  Other Names: Otezla
  Arms: Arm 1 - Standard of Care; Arm 2 - Reminder text
Behavioral: Extended Consultation for apremilast — Participants will be given their medication with the electronic adapter cap on it and will receive an initial patient consult intervention, which will focus on medication education and setting expectations of what to anticipate with usage of the prescribed medication
  Other Names: Otezla
  Arms: Arm 1 - Standard of Care; Arm 3 - Initial patient consult

SUMMARY:
Most people with psoriasis have very limited disease, yet that disease may still have a large impact on their lives. While limited psoriasis may be amenable to topical treatment, patients are exceptionally poorly adherent to topical treatment, especially over the long run.

DETAILED DESCRIPTION:
Psoriasis patients prefer oral treatments and are more adherent to orals than to topicals, but adherence to oral treatment of psoriasis may still be limited, compromising treatment outcomes. How well the medication works in the patients who take treatment regularly is not well characterized.

ELIGIBILITY:
Inclusion Criteria:

* Adult 18 years or older
* Diagnosis of mild psoriasis with Otezla recommendation
* Non-pregnant
* English speaking

Exclusion Criteria:

* Under 18 years of age
* Not diagnosis of mild psoriasis
* Pregnant
* Non-English speaking

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-06 (Estimated); Primary Completion 2025-11 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Medication Adherence Outlier | Month 6
  Identify adherence outliers (high and low adherence). Adherence will be determined by the data retrieved from the electronic monitor that is placed on the medication bottle to provide the days and times the bottle is opened to take the medication.

SECONDARY OUTCOMES:
Difference of Efficacy among high adherent subjects | Month 6
  As a secondary outcome, we will compare psoriasis treatment outcomes (efficacy) between the most and least adherent patients. Measures for comparing efficacy between high vs low adherence subjects will be percent of subjects with Investigator Global Assessment (IGA) of clear/almost clear - The IGA is a five-point scale that provides a global clinical assessment of Atopic Dermatitis (AD) severity ranging from 0 to 4, where 0 indicates clear, 2 is mild, 3 is moderate, and 4 indicates severe Atopic Dermatitis (AD). A decrease in score relates to an improvement in signs and symptoms.
Difference of Safety among low adherent subjects | Month 6
  As a secondary outcome, we will compare psoriasis treatment outcomes (safety) between the most and least adherent patients. Measures for comparing safety between high vs low adherence subjects will be percent of subjects with Investigator Global Assessment (IGA) of clear/almost clear - The IGA is a five-point scale that provides a global clinical assessment of Atopic Dermatitis (AD) severity ranging from 0 to 4, where 0 indicates clear, 2 is mild, 3 is moderate, and 4 indicates severe Atopic Dermatitis (AD). A decrease in score relates to an improvement in signs and symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Steven R Feldman, MD, PhD, Principal Investigator — Wake Forest University Health Science
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

REFERENCES:
- [Background] Salisbury KR, Ranpariya VK, Feldman SR. Accountability in reminder-based adherence interventions: A review. Patient Educ Couns. 2022 Aug;105(8):2645-2652. doi: 10.1016/j.pec.2021.12.009. Epub 2021 Dec 15. PMID 34953618
- [Background] Okwundu N, Cardwell LA, Cline AE, Richardson IM, Feldman SR. Adherence to topical treatment can improve treatment-resistant moderate psoriasis. Cutis. 2020 Feb;105(2):89-91;E2;E3. PMID 32186523
- [Background] Alinia H, Moradi Tuchayi S, Smith JA, Richardson IM, Bahrami N, Jaros SC, Sandoval LF, Farhangian ME, Anderson KL, Huang KE, Feldman SR. Long-term adherence to topical psoriasis treatment can be abysmal: a 1-year randomized intervention study using objective electronic adherence monitoring. Br J Dermatol. 2017 Mar;176(3):759-764. doi: 10.1111/bjd.15085. Epub 2016 Nov 29. PMID 27664969
- [Background] West C, Narahari S, O'Neill J, Davis S, Huynh M, Clark A, Boles A, Feldman SR. Adherence to adalimumab in patients with moderate to severe psoriasis. Dermatol Online J. 2013 May 15;19(5):18182. PMID 24011280
- [Background] Yentzer BA, Wood AA, Sagransky MJ, O'Neill JL, Clark AR, Williams LL, Feldman SR. An Internet-based survey and improvement of acne treatment outcomes. Arch Dermatol. 2011 Oct;147(10):1223-4. doi: 10.1001/archdermatol.2011.277. No abstract available. PMID 22006146